CLINICAL TRIAL: NCT03017365
Title: Effects of Different Resistance Training Methods on Strength, Motor Control and Executive Functions in Older Adults
Brief Title: Effects Resistance Training on Motor Control and Cognition
Acronym: KFPS_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kassel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFPS17
Record Dates: First submitted 2017-01-04; First posted 2017-01-11 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Muscle Weakness
Keywords: Motor Control; Balance
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- M-SRT (Active Comparator): Machine-based stable resistance training. Exercising 'traditional' machine-based resistance training.
  Interventions: Other: Stable Resistance Training
- F-URT (Experimental): Free weight unstable resistance training; conducted free-weight resistance training on unstable devices using dumbbells instead of exercise-machines.
  Interventions: Other: Unstable Resistance Training
- M-ART (Experimental): Machine-based adductor/abductor resistance training. Exercising with 'traditional' adductor/abductor machines.
  Interventions: Other: Adductor/Abductor Resistance Training

INTERVENTIONS:
Other: Stable Resistance Training — traditional machine-based resistance training
  Arms: M-SRT
Other: Unstable Resistance Training — free weight resistance training using unstable devices
  Arms: F-URT
Other: Adductor/Abductor Resistance Training — machine-based adductor/abductor resistance training
  Arms: M-ART

SUMMARY:
It is well documented that both balance and resistance training have the potential to mitigate intrinsic fall risk factors in older adults. Recently, it was shown that a simultaneously executed balance and resistance training, namely resistance training on uneven surfaces is an eligible, effective and safe alternative training program to mitigate intrinsic fall risk factors in older adults. However, knowledge about the effects of specific adductor and abductor training has advantages over traditional resistance training and resistance training on unstable surfaces regarding forward propulsion. Further, the effects of different kinds of resistance training on cognition, especially embodiment is investigated.

DETAILED DESCRIPTION:
Introduction: In the course of ageing, physical abilities decline and consequently there is an increase in risk of falling and fall incidences. Notwithstanding, the fact that causes of falls are multifactorial, losses in lower-extremity muscle strength, power and balance seem to be the most prominent intrinsic (i.e., person-related) fall risk factors in older adults. Several systematic reviews and meta-analyses highlighted the positive effects of resistance and balance training when applied as a single means, on measures of leg muscle strength, power and balance in older adults. Recently, it was shown that a simultaneously executed balance and resistance training, namely resistance training on uneven surfaces is an eligible, effective and safe alternative training program to mitigate intrinsic fall risk factors in older adults. Based on several investigations, it can be safely assumed that exercises conducted on unstable devices activate smaller muscles and stabilising function of bigger muscle groups. This facilitates torque and power transfer from lower to upper extremeties and is possibly responsible for similar effects as compared to stable resistance training despite lower loads. However, it is unknown if resistance training targeting adductor and abductor muscles induces similar results as compared to resistance training conducted on uneven surfaces. Moreover, physical activity has proven to affect cognitive measures positively, especially executive functions. It has yet to be determined to what extent different kinds of resistance training affect executive functions.

Methods/Design: This study is a three-arm, 10-week RCT with a 10-week no-contact follow-up. Participants were randomly allocated (1:1) to either: 1) machine-based stable resistance training (M-SRT); 2) free-weight unstable resistance training (F-URT); 3) machine-based adductor and abductor resistance training. The design and reporting of this study follows the CONSORT (Consolidated Standards of Reporting Trials) 2010 Statement for parallel group randomised trials.

Setting Participants are recruited from the communities in and around Kassel, Germany. Screening visits, measurement sessions, and the interventions are held at the Insitute of Sports and Sports Science / University of Kassel, Germany.

Recruitment strategies: Recruitment is carried out by placing 1) an advertisement in the local newspaper, 2) during a public information meeting at the local town hall and 3) word of mouth. Interested individuals contact the study coordinator by phone, where they are provided with a brief description of the study. If responses suggest study eligibility then interested individuals are invited to attend a formal in-person screening visit.

Participants:Older adults are eligible if they: 1) are aged between 65 and 80 years old 2) and able to walk independently for more than 10m. An a priori power analysis using G*Power 3.1 with an assumed type I error of .05 and a type II error of .10 (90% statistical power, correlation among groups: .5, nonsphericity correction: 1) was computed to determine an appropriate sample size to detect medium (.50 ≤ d ≤ .79) interaction effects. The calculations were based on a study assessing the effects of core strength training using unstable devices on older adults. The analysis revealed the requirement of 54 participants (18 per group) to obtain medium "time x group" interaction effects. Considering the likelihood of dropouts, at least 83 participants are going to be recruited to compensate for a possible dropout rate of ~20%.

Interventions: All intervention groups train for ten weeks, twice per week on non-consecutive days for 60 minutes each. The 10-week intervention period consistes of a one week introductory phase and three major training blocks lasting three weeks each. Training intensity is progressively and individually increased over the 10-week training program by modulating load and sets for all groups and level of instability for F-URT. After week one (50 %), four (60%), and seven (70%) the training load (weight) is increased following one repetition maximum (1-RM) testing for each major exercise. M-SRT followes a 'traditional' machine-based stable resistance training program, including squats with a smith-machine and a leg press. F-URT conducts squats and front lunges on unstable devices. M-ART uses adductor and abductor strength training machines. All three intervention groups conduct a resistance training program consisting of two main exercises, a preparation and cool-down phase. Participants perform ten minutes of low-intensity stepping on a stair-walker as a brief warm-up at the beginning of each training session, followed by the resistance exercises and walking on a treadmill as cool-down. Training under unstable surface conditions, especially with additional weight, implies a certain degree of accident risk. Due to this factor, all instability exercises are observed by instructors and secured with additional aids like boxes. Training is supervised by skilled instructors at all times. For the first two weeks the participant to instructor ratio will be 5:1, thereafter 10:1.

Outcome assessment: Outcomes are measured at baseline, 10 weeks (intervention endpoint) and 20 weeks (study endpoint). Measurement sessions are conducted on one day.

Baseline data: Baseline measurements are obtained prior to randomisation. In addition to the measurements described below, the following are also collected: demographic and general health characteristics; medical history and medications; anthropometrics and rate of falls / near falls.

ELIGIBILITY:
Inclusion Criteria:

* between 65 and 80 years old
* ability to walk independently without any gait aid

Exclusion Criteria:

* pathological ratings of the Clock Drawing Test (CDT),
* Mini-Mental-State-Examination (MMSE, < 24 points),
* Falls Efficacy Scale - International (FES-I, > 24 points),
* Geriatric Depression Scale (GDS, > 9 points),
* Freiburg Questionnaire of Physical Activity (FQoPA, < 1hour)
* Frontal Assessment Battery (FAB-D, < 18 points)
* any neurological, musculoskeletal or heart-related disease

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Clinical Gait Analysis | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  changes in variance components (Vucm, Vort, Vtot) of an uncontrolled manifold analysis; measured in rad²

SECONDARY OUTCOMES:
Maximal isometric leg extension strength (ILES) | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in isometric strength, measured in N
Fall self-efficacy Questionnaire | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in anxiety score
Proactivec Balance (timed up and go test) | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in leg strength and procative balance (seconds)
Maximal isometric adductor and abductor strength | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in isometric strength, measured in N
Stroop Task | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in reaction time to congruent and incongruent stimuli (ms)
Proactivec Balance (multidirectional reach test) | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in proactive balance (cm)
Power tests (chair rise test) | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in muscle power (seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Armin Kibele, PhD, Study Chair — University of Kassel

IPD SHARING:
Plan to Share IPD: Yes
Raw results will be published. Age will be described as intervals (65-69, 70-74, 75-80) and height will be removed, thus no backtracking is possible
Supporting Information: SAP
Time Frame: when the article is published
Access Criteria: IPD will be published as supplementary material. Raw results will be published. Age will be described as intervals (65-69, 70-74, 75-80) and height will be removed, thus no backtracking is possible

REFERENCES:
- [Background] Eckardt N. Lower-extremity resistance training on unstable surfaces improves proxies of muscle strength, power and balance in healthy older adults: a randomised control trial. BMC Geriatr. 2016 Nov 24;16(1):191. doi: 10.1186/s12877-016-0366-3. PMID 27881086
- [Background] Granacher U, Muehlbauer T, Gruber M. A qualitative review of balance and strength performance in healthy older adults: impact for testing and training. J Aging Res. 2012;2012:708905. doi: 10.1155/2012/708905. Epub 2012 Jan 23. PMID 22315687
- [Background] Steadman J, Donaldson N, Kalra L. A randomized controlled trial of an enhanced balance training program to improve mobility and reduce falls in elderly patients. J Am Geriatr Soc. 2003 Jun;51(6):847-52. doi: 10.1046/j.1365-2389.2003.51268.x. PMID 12757574
- [Background] Behm DG, Muehlbauer T, Kibele A, Granacher U. Effects of Strength Training Using Unstable Surfaces on Strength, Power and Balance Performance Across the Lifespan: A Systematic Review and Meta-analysis. Sports Med. 2015 Dec;45(12):1645-69. doi: 10.1007/s40279-015-0384-x. PMID 26359066
- [Derived] Eckardt N, Rosenblatt NJ. Instability Resistance Training Decreases Motor Noise During Challenging Walking Tasks in Older Adults: A 10-Week Double-Blinded RCT. Front Aging Neurosci. 2019 Feb 27;11:32. doi: 10.3389/fnagi.2019.00032. eCollection 2019. PMID 30873017